CLINICAL TRIAL: NCT00290043
Title: Glucodynamic Response to Pre- and Postmeal Subcutaneous Injection of 0.15 IU/kg HMR1964 Insulin and RHI in Type 1 Diabetic Subjects in an Open, Randomized, Four-way Crossover Study
Brief Title: Glulisine Pre- and Postmeal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A/1008; HMR1964
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Insulin glulisine; Diabetes mellitus Type 1; Postprandial Period; Pharmacokinetics; Glucodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin glulisine

SUMMARY:
To investigate in type 1 diabetic patients the glucodynamic response to HMR1964 insulin and RHI (HOE31HPR100) injected subcutaneously before and after a standard meal

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-12; Study Completion 2002-03

PRIMARY OUTCOMES:
Outcome measures: Post-prandial glucose and insulin concentrations. Outcome: In T1DM, insulin glulisine provides a better mimic of the physiological postprandial glucose disposal than RHI.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Rave, Dr., Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com